CLINICAL TRIAL: NCT01981356
Title: Acceptance and Commitment Therapy for the Inpatient Treatment of Psychosis
Acronym: ACT-IP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPO 13-132
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Psychotic Disorders
Keywords: Psychotic Disorders; Acceptance and Commitment Therapy; Inpatient psychiatry; Schizophrenia; Acute psychiatric disorder
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Acceptance and Commitment Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acceptance and Commitment Therapy (ACT) (Experimental): Participants randomized to the ACT condition will be provided with the opportunity to attend 4 ACT sessions. The treatment protocol is adapted from and virtually identical to that presented in Gaudiano and Herbert (2006). Each ACT session will serve as a standalone session, with all essential elements of the treatment briefly presented. Participants in the ACT condition will also receive treatment as usual.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Treatment as Usual (TAU) (Active Comparator): TAU consists of psychopharmacology, case management, and psychotherapy. Additionally, patients randomized to the TAU condition will meet with ACT facilitators for 15 minutes every other day to provide additional support and answer questions, while ensuring not to discuss or suggest the use of therapeutic techniques related to ACT.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — The goal of ACT is to help the patient increase psychological flexibility, a core component of mental health and well-being. ACT teaches clients to be mindfully aware but nonreactive to delusions/ hallucinations and to increase willingness to
  experience associated distressing emotions while simultaneously engaging in meaningful behavioral actions.
  Patients expand their repertoire of behaviors to live according to their values and to pursue valued goals, thereby increasing adaptive functioning and quality of life.
  Other Names: ACT
  Arms: Acceptance and Commitment Therapy (ACT)
Other: Treatment as Usual (TAU) — All patients admitted to the acute psychiatry unit are administered anti-psychotic and/or other psychotropic medication during their inpatient stay. Patients participate in standard milieu therapy on the unit (group and activities therapies, and individual therapy as needed). Therapy on the unit focuses on psycho-education about illness, symptom identification, mood management techniques, stress reduction, and relapse prevention. Patients also receive unstructured individual therapy and case management as appropriate.
  Arms: Treatment as Usual (TAU)

SUMMARY:
There is a substantial need for enhancing the efficacy and effectiveness of Veterans Health Administration (VHA) inpatient services for psychosis and tailoring them to support recovery. The proposed pilot study will explore whether Acceptance and Commitment Therapy (ACT), a recovery-oriented, evidence-based inpatient treatment, is a feasible, acceptable, safe, and effective adjunct for the inpatient treatment of Veterans with psychosis at a single VHA site. Additionally, an evaluation of barriers and facilitators to future implementation will be conducted. If promising, the data gained from the proposed study will support future evaluation, implementation and dissemination efforts that have the potential to improve inpatient treatment for psychosis and recovery, and thus, the lives of Veterans, while reducing costs for VHA.

DETAILED DESCRIPTION:
Within the Veterans Health Administration (VHA) in fiscal year 2011, patients with psychotic disorders represented approximately 4% of the total population, and received approximately 14% of VHA's total expenditures (Blow et al., 2011). Patients with psychosis receive substantial, repeated, and costly inpatient treatment, and this is often the only chance to provide treatment due to gaps in mental health service utilization (Blow et al., 2011; McCarthy et al., 2007). Thus, there is an urgent need for enhancing the efficacy and effectiveness of VHA inpatient services and tailoring them to better support recovery.

Acceptance and Commitment Therapy (ACT), a recovery-oriented, evidence-based adjunct to inpatient treatment for psychosis, is an excellent candidate for investigations within VHA inpatient settings. ACT for psychosis is considered an empirically supported treatment by the American Psychological Association (APA, 2012; Chambless et al., 1998). A consistent body of research has demonstrated the clinical effectiveness of ACT for treatment of psychosis, including well-designed randomized clinical trials of ACT on inpatient settings (Bach & Hayes, 2000; Gaudiano & Herbert, 2006). ACT is effective when provided in a flexible format of three to four sessions, and for patients with a range of chronic and severe psychotic and comorbid mental disorders.

This proposed pilot study aims to explore ACT as an adjunct to inpatient treatment as usual (TAU) for psychosis among VHA patients at one VHA inpatient psychiatry unit. The project will use an effectiveness/ implementation Hybrid Type 1 design that incorporates a pilot RCT and semi-formative evaluation of barriers and facilitators to future implementation. Participants will be 80 VHA patients with current psychotic symptoms (hallucinations and/or delusions) related to a psychotic or mood disorder who are admitted to an inpatient psychiatry unit VA Palo Alto Health Care System (VAPAHCS). Participants will be randomly assigned to receive either TAU (n = 40), or TAU with plus 4-sessions of ACT (n = 40) individually provided during their stay on the inpatient unit. Aim 1 is to investigate the feasibility, acceptability, and safety of the treatment for VHA patients, as indexed by: (a) the ability to recruit and consent 2 eligible participants per week (for 40 weeks) to participate in the study and be randomized to ACT + TAU or TAU; (b) patient attendance of 3 ACT individual sessions (out of 4 possible) on average; (c) patient and ACT Facilitator (provider of the intervention), reported ACT treatment satisfaction and alliance; and (d) the occurrence of zero serious adverse events attributable to the ACT treatment. Aim 2 is to investigate treatment effects of ACT on patient functioning (i.e., acceptance), symptomatology, distress, and affect. Aim 3 is to obtain data from participating patients and unit staff regarding system-, clinician- and patient-level barriers and facilitators to implementing staff-delivered ACT services for psychosis at the participating VHA inpatient setting, including: (a) barriers that limit patients, staff, and site participation in ACT and how to address them; (b) provider and patient perceptions about why ACT is successful at achieving better outcomes; (c) site specific and general barriers to implementation of ACT and how to address them; and (d) perceived value of and how to sustain ACT in the absence of a funded project.

This project is the first step in exploring a potentially sustainable and effective intervention that will improve inpatient psychosis treatment and recovery, and hence, the lives of VHA patients with psychosis, while reducing costs for VHA. If promising, study findings will support a HSR&D Investigator Initiated Research (IIR) Merit grant application that will propose to assess the effectiveness and cost of implementing the ACT intervention, and potential barriers and facilitators for implementation efforts at multiple VHA inpatient psychiatric units. The aims of this project align with the HSR&D research priority area of improving mental and behavioral interventions for individuals with serious mental illness by refining recovery-oriented treatment approaches related to evidence-based programs.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the patient sample, used to establish feasibility, acceptability, safety, and efficacy of the experimental treatment, will be:

* hospitalized with current psychosis symptoms (hallucinations and/or delusions);
* DSM-IV-TR (APA, 2000) diagnosis of a psychotic disorder (i.e., schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, brief psychotic disorder, psychotic disorder not otherwise specified) or a mood disorder with psychotic features (major depression, bipolar I disorder) that requires hospitalization;
* ability to provide informed consent ;
* conversational in English; and
* patient stay on the unit estimated in advance to be greater than one week.

Inclusion criteria for the staff sample, used to identify barriers and facilitators to the implementation of the experimental treatment, will be

* ability to provide informed consent and
* conversational in English.

Exclusion Criteria:

None.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T Boden, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We reviewed charts for 429 admissions over 8 months; 67 patients were approached because they potentially met study criteria
Pre-assignment Details: Although 18 participants were randomized to treatment condition, the consent of two participants was invalid. Thus, their data could not be utilized and is not reported other than for identification of participant flow.
Groups:
- Acceptance and Commitment Therapy (ACT): Participants randomized to the ACT condition will be provided with the opportunity to attend 4 ACT sessions, all of which will occur within 9 days of the patient's admission to the inpatient unit. Each ACT session will serve as a standalone session, with all essential elements of the treatment briefly presented. Each session will contain a core set of themes and exercises that will be rotated over subsequent sessions (e.g., acceptance of uncontrollable vs. controllable events). Each session will begin with a brief psycho-educational component to address psychotic symptoms, followed by presentation of the ACT model to provide a rationale for treatment. Participants in the ACT condition will also receive treatment as usual.
Period: Overall Study
Arm/Group | Acceptance and Commitment Therapy (ACT) | Treatment as Usual (TAU)
Started | 12 | 6
Completed | 5 | 4
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: Although 18 participants were randomized to treatment condition, the consent of two participants was invalid. Thus, their data could not be utilized and is not reported other than for identification of participant flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acceptance and Commitment Therapy (ACT) | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (16.2) | 55.8 (17.7) | 53.7 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 6 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 4 | 2 | 6
  Hispanic or Latino/a | 2 | 2 | 4
  Black or African American | 2 | 2 | 4
  Asian or Asian American | 1 | 0 | 1
  Not reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Brief Psychiatric Rating Scale (Overall & Gorham, 1962)
Description: Assesses changes in broad symptom domains (affect disturbance, positive symptoms, negative symptoms, resistance/hostility, activation) and specific symptoms (e.g., delusions). All scale items were averaged to obtain a total scale score. Scale scores are reported as percentage of total possible change, calculated as follow-up score minus baseline score divided by total points in scale. Minimum score is -100% change (a decrease of 100% of total possible score from baseline to follow-up assessment). Minimum score is akin to a change from the highest (7) to lowest (1) possible value on scale from baseline to follow-up. Maximum score is +100% change (an increase of 100% of total possible score from baseline to follow-up assessment). Maximum score is akin to a change from the lowest (1) to highest (7) possible value on scale from baseline to follow-up. Decreases in percentage change are considered better outcomes (i.e., reduced symptoms).
Time Frame: Participants were followed for the duration of hospital stay (Mean = 24.0 days, SD = 15.8).
Measure: Mean (Standard Deviation); unit: percentage of total possible change
Arm/Group | Acceptance and Commitment Therapy (ACT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 5 | 4
percentage of total possible change | -8.0 (13.8) | -11.6 (5.8)

2. Secondary Outcome: Frequency, Believability, and Distress Symptom Scale (Gaudiano & Herbert, 2006)
Description: Assesses changes in the frequency, believability, and associated distress of psychosis symptoms. Frequency, believability, and distress subscales consist of two items each, one assessing delusions and one assessing hallucinations, averaged to obtain subscale scores. Subscale scores are reported as percentage of total possible change, calculated as follow-up score minus baseline score divided by total points in scale. Minimum score is -100% change (a decrease of 100% of total possible score from baseline to follow-up assessment). Minimum score is akin to a change from the highest to lowest possible value on scale from baseline to follow-up. Maximum score is +100% change (an increase of 100% of total possible score from baseline to follow-up assessment). Maximum score is akin to a change from the lowest to highest possible value on scale from baseline to follow-up. Decreases in percentage change are considered better outcomes (i.e., reduced frequency, believability and distress).
Time Frame: Participants were followed for the duration of hospital stay (Mean = 24.0 days, SD = 15.8).
Population: Out of participants who completed follow-up assessments, one participant in each condition did not complete the Frequency, Believability, and Distress Symptom Scale.
Measure: Mean (Standard Deviation); unit: percentage of total possible change
Arm/Group | Acceptance and Commitment Therapy (ACT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 4 | 3
percentage of total possible change
  Frequency | -14.6 (17.2) | -22.2 (25.5)
  Believability | -15.3 (15.3) | -35.2 (61.4)
  Distress | -12.5 (14.6) | -34.7 (48.5)

3. Secondary Outcome: Acceptance and Action Questionnaire - II (Bond et al.., 2011)
Description: Assesses changes in the primary mechanism thought to contribute to change in ACT: acceptance. All scale items were averaged to obtain a total scale score. Total scale scores are reported as percentage of total possible change, calculated as follow-up score minus baseline score divided by total points in scale. Minimum score is -100% change (a decrease of 100% of total possible score from baseline to follow-up assessment). Minimum score is akin to a change from the highest (7) to lowest (1) possible value on scale from baseline to follow-up. Maximum score is +100% change (an increase of 100% of total possible score from baseline to follow-up assessment). Maximum score is akin to a change from the lowest (1) to highest (7) possible value on scale from baseline to follow-up. Increases in percentage change are considered better outcomes (i.e., increased acceptance).
Time Frame: Participants were followed for the duration of hospital stay (Mean = 24.0 days, SD = 15.8).
Population: Out of participants who completed follow-up assessments, one participant in each condition did not complete the Acceptance and Action Questionnaire - II.
Measure: Mean (Standard Deviation); unit: percentage of total possible change
Arm/Group | Acceptance and Commitment Therapy (ACT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 4 | 3
percentage of total possible change | 14.5 (29.6) | 19.8 (33.9)

4. Secondary Outcome: Positive and Negative Affect Scale (Watson et al., 1988)
Description: Assesses short-term changes in global positive and negative affect in addition to changes in specific types of emotions (e.g., afraid, excited, guilty). Positive and negative affect subscales consist of ten items each, averaged to obtain scale scores. Scale scores are reported as percentage of total possible change, calculated as follow-up score minus baseline score divided by total points in scale. Minimum score is -100% change (a decrease of 100% of total possible score from baseline to follow-up assessment). Minimum score is akin to a change from the highest (5) to lowest (1) possible value on scale from baseline to follow-up. Maximum score is +100% change (an increase of 100% of total possible score from baseline to follow-up assessment). Maximum score is akin to a change from the lowest (1) to highest (5) possible value on scale from baseline to follow-up. Increases in positive affect percentage change and decreases in negative affect change are considered better outcomes.
Time Frame: Participants were followed for the duration of hospital stay (Mean = 24.0 days, SD = 15.8).
Measure: Mean (Standard Deviation); unit: percentage of total possible change
Arm/Group | Acceptance and Commitment Therapy (ACT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 5 | 4
percentage of total possible change
  Positive Affect | 16.5 (37.0) | 18.1 (32.5)
  Negative Affect | -15.5 (30.9) | -27.5 (40.6)

5. Secondary Outcome: Cost of Stay
Description: Obtained by: (a) obtaining length obtained by: (a) obtaining length-of-stay (in hours) on the inpatient unit for all study participants, (b) calculating the cost of stay for each participant by multiplying the length-of-stay by the dollar amount associated with inpatient treatment of psychosis (e.g., $1,297/day or $54/hour in 2011; Blow et al., 2011), and (c) summing the cost of stay across participants in each treatment condition.
Time Frame: Participants were followed for the duration of hospital stay (Mean = 24.0 days, SD = 15.8).
Population: Data regarding length of stay not available for one participant in each condition, both of whom had not been discharged by the end of the study period.
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Acceptance and Commitment Therapy (ACT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 4 | 3
Dollars | 43,728.75 (26,190.96) | 25,415.00 (19,086.88)

6. Secondary Outcome: Barriers and Facilitators to Implementation
Description: We will conduct 30-60 minute semi-structured interviews structured around the RE-AIM framework (Glasgow et al., 1999), and utilizing the RE-AIM Planning Tool (Forman et al., 2010). The RE-AIM framework identifies, for example, barriers that limit patients, staff, and site participation in the intervention and how to address them, and provider and patient perceptions about why the intervention is successful at achieving better outcomes.
Time Frame: 8-month study period
Population: Data regarding barriers and facilitators was not obtained from patient participants, but was obtained from study staff, who were not assigned to treatment condition.
Measure: Number; unit: Participants providing data
Groups:
- Inpatient Psychiatry Unit Staff Members: Barriers and facilitators were assessed through interviews of four inpatient psychiatry unit staff (on nursing assistant, one nurse, two psychologists).
Arm/Group | Inpatient Psychiatry Unit Staff Members
Number analyzed (Participants) | 4
Participants providing data | 4

7. Secondary Outcome: Experimental Treatment Feasibility
Description: Assessed by our ability to recruit and consent 2 eligible participants per week (for 40 weeks) to participate in random assignment to ACT + TAU or TAU.
Time Frame: 8-month study period
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Acceptance and Commitment Therapy (ACT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 6
participants | 10 | 6

8. Secondary Outcome: Experimental Treatment Acceptability
Description: Assessed by patient attendance of at least 3 out of 4 sessions on average.
Time Frame: 8-month study period
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Acceptance and Commitment Therapy (ACT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 5 | 4
sessions | 4.0 (0.0) | 3.5 (1.0)

9. Secondary Outcome: Experimental Treatment Safety
Description: Assessed by the occurrence of zero adverse events attributable to ACT.
Time Frame: 8-month study period
Population: as for baseline characteristics
Measure: Number; unit: adverse events
Arm/Group | Acceptance and Commitment Therapy (ACT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 6
adverse events | 0 | 0

10. Secondary Outcome: Experimental Treatment Acceptability
Description: Assessed by patient reported treatment satisfaction, as assessed by the well-validated Client Satisfaction Questionnaire - 8 (CSQ-8; Attkisson & Zwick, 1982; range 0 to 5, higher scores indicate better outcome).
Time Frame: Participants were followed for the duration of hospital stay (Mean = 24.0 days, SD = 15.8).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance and Commitment Therapy (ACT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 5 | 4
units on a scale | 2.9 (0.3) | 3.3 (0.4)

11. Secondary Outcome: Experimental Treatment Acceptability
Description: Assessed by patient reported therapeutic alliance, measured by the well-validated Working Alliance Inventory (WAI; Horvath & Greenberg, 1989; range 1 to 7, higher score indicated better outcome).
Time Frame: Participants were followed for the duration of hospital stay (Mean = 24.0 days, SD = 15.8).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance and Commitment Therapy (ACT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 5 | 4
units on a scale | 4.7 (1.0) | 5.3 (1.1)

ADVERSE EVENTS:
Time Frame: 8 months
Description: Time frame for adverse event reporting is from the beginning to the end of the trial.
Arm/Group | Acceptance and Commitment Therapy (ACT) | Treatment as Usual (TAU)
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 0/12 | 0/6

LIMITATIONS AND CAVEATS:
Patient recruitment was hindered by patient characteristics, and inherent difficulties in conducting research with psychiatry inpatients. These issues do not address whether ACT is a beneficial inpatient treatment for psychosis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes